CLINICAL TRIAL: NCT04676139
Title: The Safety and Efficacy of Selective Serotonin Reuptake Inhibitors, Fluoxetine, for Refractory Primary Mono-symptomatic Nocturnal Enuresis in Children: A Randomized Controlled Trial
Brief Title: The Safety and Efficacy of Fluoxetine for Refractory Primary Mono-symptomatic Nocturnal Enuresis in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSRI & Nocturnal enuresis
Record Dates: First submitted 2020-12-05; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine (Experimental): patients will undergo maintenance therapy selective serotonin reuptake inhibitors, fluoxetine, 10 mg capsules once daily for 12 weeks
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): patients will undergo maintenance therapy Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 10 mg capsules once daily for 12 months
  Arms: Fluoxetine
Drug: Placebo — placebo for 12 months
  Arms: Placebo

SUMMARY:
To determine whether there is a role for the selective serotonin reuptake inhibitors, fluoxetine, as therapy in the treatment of refractory primary monosymptomatic nocturnal enuresis in children , and whether there are side effects involved.

ELIGIBILITY:
Inclusion Criteria:

* Primary Monosymptomatic nocturnal enuresis
* Failed treatment with desmopressin.
* The enuresis alarm had either been tried without effect, or deemed unfeasible because of the family situation.
* All patients had either tried and failed combination therapy with anticholinergics or, because of contraindications, been unable to receive such therapy.
* Severe enuresis with at least seven wet nights out of 14

Exclusion Criteria:

* Underlying renal, urologic, neurologic, endocrinologic, or cardiac conditions
* Depression
* Severe psychiatric diseases
* Untreated constipation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
assess efficacy Selective Serotonin Reuptake Inhibitors, Fluoxetine, for refractory Primary Mono-symptomatic Nocturnal Enuresis in children. | 6 months
  counting the wet nights numbers between baseline and after 2 weeks of each treatment period

SECONDARY OUTCOMES:
assess the safety of Selective Serotonin Reuptake Inhibitors, Fluoxetine, for refractory Primary Mono-symptomatic Nocturnal Enuresis in children. | 6 months
  by counting the numbers of complication of each drugs

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkenawy, Study Chair — Professor of urology Urology and Nephrology center Faculty of medicine Mansoura university; Tamer El-sayed Helmy, Study Director — Associate Professor of urology Urology and Nephrology center Faculty of medicine Mansoura university; Ahmed Abdelhalem, Study Director — Lecturer of urology Urology and Nephrology center Faculty of medicine Mansoura university; Mohamed Hussiny abdelazim, Principal Investigator — Resident in Urology Urology and Nephrology canter Mansoura University
Locations (1):
- Mansoura urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neveus T. Pathogenesis of enuresis: Towards a new understanding. Int J Urol. 2017 Mar;24(3):174-182. doi: 10.1111/iju.13310. Epub 2017 Feb 16. PMID 28208214
- [Result] Neveus T, Eggert P, Evans J, Macedo A, Rittig S, Tekgul S, Vande Walle J, Yeung CK, Robson L; International Children's Continence Society. Evaluation of and treatment for monosymptomatic enuresis: a standardization document from the International Children's Continence Society. J Urol. 2010 Feb;183(2):441-7. doi: 10.1016/j.juro.2009.10.043. Epub 2009 Dec 14. PMID 20006865
- [Result] Song P, Huang C, Wang Y, Wang Q, Zhu W, Yue Y, Wang W, Feng J, He X, Cui L, Wan T, Wen J. Comparison of desmopressin, alarm, desmopressin plus alarm, and desmopressin plus anticholinergic agents in the management of paediatric monosymptomatic nocturnal enuresis: a network meta-analysis. BJU Int. 2019 Mar;123(3):388-400. doi: 10.1111/bju.14539. Epub 2018 Oct 31. PMID 30216627